CLINICAL TRIAL: NCT00603473
Title: An Open-Label, Multicenter Study Evaluating, The Efficacy, Safety And Pharmacokinetics Of Gabapentin As Adjunctive Therapy In Pediatric Patients With Partial Seizures When Other Antiepileptics Do Not Provide Satisfactory Effects
Brief Title: A Phase III Open-Label Study Of Gabapentin As Adjunctive Therapy In Japanese Pediatric Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9451162
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2011-01

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gabapentin (Experimental)
  Interventions: Drug: gabapentin

INTERVENTIONS:
Drug: gabapentin — Orally administered gabapentin

SUMMARY:
Examine the efficacy, safety and pharmacokinetics of gabapentin as adjunctive therapy in Japanese pediatric patients with partial seizures

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or females, ages 3-15 years old at acquisition of informed consent, 15 years old or less at the baseline visit
* Seizures are classified as simple partial, complex partial or partial becoming secondarily generalized (defined according to the International League Against Epilepsy)
* Have not been able to achieve adequate seizure control with antiepileptic drugs

Exclusion Criteria:

* Seizures related to drugs or acute medical illness
* History of any serious medical or psychiatric disorder
* Diagnosis or history of a structural CNS lesion or an encephalopathy shown to be progressive

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- Japan (26):
  - Pfizer Investigational Site, Obu-shi,Morioka-machi, Aichi-ken
  - Pfizer Investigational Site, Jonan-ku, Fukuoka
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Suma-Ku, Kobe, Hyōgo
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Zentsuuji, Kagawa-ken
  - Pfizer Investigational Site, Yokohama, Kanagawa Pref.
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Shōwaku, Nagoya
  - Pfizer Investigational Site, Niigata, Niigata
  - Pfizer Investigational Site, Kurashiki, Okayama Pref.
  - Pfizer Investigational Site, Okayama, Okayama-ken
  - Pfizer Investigational Site, Izumi-shi, Osaka
  - Pfizer Investigational Site, Miyakojima-ku, Osaka
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Higashi-Matsuyama, Saitama
  - Pfizer Investigational Site, Shizuoka, Shizuoka
  - Pfizer Investigational Site, Kiyose-shi, Tokyo
  - Pfizer Investigational Site, Kodaira, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Hiroshima
  - Pfizer Investigational Site, Saitama
  - Pfizer Investigational Site, Yamagata
  - Pfizer Investigational Site, Yamanashi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451162&StudyName=A%20Phase%20III%20Open-Label%20Study%20Of%20Gabapentin%20As%20Adjunctive%20Therapy%20In%20Japanese%20Pediatric%20Patients%20With%20Partial%20Seizures

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 27 centers in Japan.
Pre-assignment Details: Ninety subjects were enrolled in the study. Of them, 89 received the study treatment, while 1 withdrew consent.
Groups:
- Gabapentin: The dosage of oral solution for subjects aged 3 to 12 years was calculated based on their body weight. The dose was titrated for the first 3 days of the treatment period. Subjects aged 3 to 4 years received gabapentin 10 mg/kg/day on Day 1, 20 mg/kg/day on Day 2 and 40 mg/kg/day from Day 3. Subjects aged 5 to 12 years received gabapentin 10 mg/kg/day on Day 1, 20 mg/kg/day on Day 2 and 25 to 35 mg/kg/day from Day 3. Subjects aged 13 to 15 years received gabapentin 600 mg/day on Day 1, 1200 mg/day on Day 2 and 1200 or 1800 mg/day from Day 3. After Day 3, the dose was adjusted if necessary within the range of maintenance doses. The maximum daily dose was 600 mg for Day 1, 1200 mg for Day 2, and 1800 mg for Day 3 and thereafter.
Period: Overall Study
Arm/Group | Gabapentin
Started | 89
Completed | 80
Not Completed | 9
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 4
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gabapentin
Number analyzed (Participants) | 89
Age, Customized [Number; unit: Subjects]
  >= 3 years and < 5 years | 11
  >= 5 years and < 13 years | 63
  >= 13 years and =< 15 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Response Ratio of Gabapentin in Japanese Pediatric Patients With Partial Seizures
Description: The Response Ratio calculated by the following equation was assessed as the primary endpoint: R Ratio = (T-B) / (T+B) where T is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 12-week treatment period, and B is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 6-week baseline period.
Time Frame: 12 weeks
Population: Modified intent-to-treat (MITT) population: Subjects who have received the study medication for at least 28 days and in whom the number of epileptic seizures used for efficacy assessment has been counted for at least 28 days in both the baseline and treatment periods.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Gabapentin
Number analyzed (Participants) | 86
ratio | -0.158 [-0.221 to -0.096]

2. Secondary Outcome: Responder Rate
Description: Responder Rate was defined as the percentage of subjects with a 50% or greater reduction in the seizure frequency per 28 days for the 12-week treatment period in comparison with the frequency per 28 days for the 6-week baseline period.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Gabapentin
Number analyzed (Participants) | 86
Percentage of Subjects | 19.8 [12.0 to 29.8]

3. Secondary Outcome: Percent Change in Seizure Frequency (PCH)
Description: PCH calculated by the following equation was assessed as secondary endpoint: PCH = 100 (T-B) / B where T is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 12-week treatment period, and B is seizure frequency per 28 days (i.e., the number of seizures per 28 days) calculated from the total number of seizures for the 6-week baseline period.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Gabapentin
Number analyzed (Participants) | 86
Percent Change | -24.4 [-100.0 to 192.9]

ADVERSE EVENTS:
Time Frame: 12-week treatment period, and 1-week follow-up period
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Gabapentin
Serious Adverse Events (participants affected / at risk) | 1/89
Other Adverse Events (participants affected / at risk) | 73/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=89)
Pharyngitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=89)
Conjunctivitis (Eye disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 5
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 24
Pharyngitis (Infections and infestations) | 6
Rhinitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 6
Excoriation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 7
Increased appetite (Metabolism and nutrition disorders) | 3
Ataxia (Nervous system disorders) | 3
Convulsion (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 35
Rash (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.